CLINICAL TRIAL: NCT04960449
Title: Arthroscopic Treatment of Partial-thickness Rotator Cuff Tendon Tears
Brief Title: Arthroscopic Treatment of Partial Rotator Cuff Tears in Shoulder Joint
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2014101
Record Dates: First submitted 2021-06-27; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-06

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with partial-thickness rotator cuff tendon tears: Partial rotator cuff tears can be divided into three categories, bursa side tears, tendon tears and joint side tears. Studies have found that rotator cuff tendon tears account for 55% of partial tears, compared to the other two types of partial tears, there has been very little research on partial-thickness rotator cuff tendon tears, which has no consensus on diagnosis and treatment.
  Interventions: Procedure: shoulder arthroscopy

INTERVENTIONS:
Procedure: shoulder arthroscopy — Patients underwent ubacromial bursectomy and acromioplasty , cuff debridement and cuff repair, side to side suture of rotator cuff combined with suture anchor.

SUMMARY:
A retrospective analysis was performed on patients with partial-thickness rotator cuff tendon tears who underwent arthroscopic surgery from August 2006 to December 2011. To evaluate functional outcomes and tendon healing after arthroscopy.

DETAILED DESCRIPTION:
To study the surgical method and clinical effect of arthroscopic treatment of rotator cuff tendon tear. Retrospective analysis was performed on patients with rotator cuff tendon tears who underwent arthroscopic surgery from August 2006 to December 2011. Preoperative X-ray and MRI were performed. Rotator cuff repair was performed during the operation. UCLA shoulder scoring scale was used to evaluate the shoulder joint at preoperative and final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* From August 2006 to December 2011, patients with partial-thickness rotator cuff tendon tears who underwent arthroscopic surgery in our department and were successfully followed up.

Exclusion Criteria:

* Patients with frozen shoulder and shoulder joint instability.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with partial-thickness rotator cuff tendon tears. Partial rotator cuff tears can be divided into three categories, bursa side tears, tendon tears and joint side tears. Studies have found that rotator cuff tendon tears account for 55% of partial tears, compared to the other two types of partial tears, there has been very little research on partial-thickness rotator cuff tendon tears, which has no consensus on diagnosis and treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
The function of shoulder joint was analyzed 1 year after arthroscopy. | 1 year after operation
  The range of motion and strength of the shoulder joint in all directions are evaluated and recorded. Analysis of UCLA (University of California, Los Angeles) Shoulder Score Scale at 1 year after operation.The UCLA scale has a minimum score of 2 and a maximum score of 35. The higher the score, the better the prognosis of the patients.
The function of shoulder joint was analyzed 2 years after arthroscopy. | 2 years after operation
  The range of motion and strength of the shoulder joint in all directions are evaluated and recorded. Analysis of UCLA Shoulder Score Scale at 2 years after operation
The function of shoulder joint was analyzed 5 years after arthroscopy. | 5 years after operation
  The range of motion and strength of the shoulder joint in all directions are evaluated and recorded. Analysis of UCLA Shoulder Score Scale at 5 years after operation

CONTACTS AND LOCATIONS:
Overall Officials: jian xiao, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No